CLINICAL TRIAL: NCT05586516
Title: A Phase 1b, Open Label, Dose Escalation Study of IOA-289, an Orally Bioavailable, Selective Autotaxin (ENPP2) Inhibitor Alone and in Combination with Gemcitabine/nab-paclitaxel in Patients with Metastatic Pancreatic Cancer
Brief Title: A Study to Assess an ATX Inhibitor (IOA-289) in Patients with Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: iOnctura (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOA-289-102
Record Dates: First submitted 2022-10-13; First posted 2022-10-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Metastatic; Pancreatic; Cancer; Autotaxin; ATX; Lysophosphatidic acid; LPA; Fibrosis; Immune
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Neoplasms; Fibrosis | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IOA-289 in combination with gemcitabine/nab-paclitaxel (Experimental)
  Interventions: Drug: IOA-289

INTERVENTIONS:
Drug: IOA-289 — IOA-289 will be administered orally twice daily (BID), starting from C0D1. Gemcitabine and nab-paclitaxel will be administrated by IV infusion, weekly for 3 weeks of a 4 week cycle starting at C1D1.
  Other Names: gemcitabine; nab-paclitaxel; Abraxane

SUMMARY:
The objective of study IOA-289-102 is to evaluate the safety and tolerability of escalating doses of IOA-289 in patients with metastatic pancreatic cancer in combination with standard chemotherapy consisting of gemcitabine and nab-paclitaxel. Blood and tumour samples for PK and PD will be collected and assessments for determination of any clinical efficacy will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age inclusive, at the time of signing the informed consent.
2. Capable of giving signed informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
4. Patients with histologically or cytologically confirmed metastatic unresectable pancreatic adenocarcinoma.
5. Have measurable disease (≥ 1 measurable lesion) based on Response Evaluation Criteria In Solid Tumours (RECIST) v1.1 as determined by the site study team.
6. Eligible to receive 1st line systemic treatment with gemcitabine/nab-paclitaxel for metastatic disease.
7. Baseline CA19-9 levels are available from a sample acquired no more than 4 weeks prior to screening.
8. No prior systemic anti-cancer therapy for metastatic pancreatic cancer.
9. Male subjects with female partners of childbearing potential, and female subjects of child-bearing potential who had a negative serum pregnancy test at screening, must agree to use a highly effective form of contraception (with at least 99% certainty) or avoid intercourse during and upon completion of the study and for at least 3 months after the last dose of study drug.

Exclusion Criteria:

1. Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications.
2. Have prior significant medical history and AEs:

   1. Known active CNS metastases and/or carcinomatous meningitis.
   2. History or presence of an abnormal ECG that, in the Investigator's opinion, is clinically meaningful. Screening QTc interval > 480 milliseconds is excluded (corrected by Fridericia).
   3. Known additional malignancy that is progressing or requires active treatment. Patients with active malignancy requiring concurrent intervention or previous malignancies (for example non-melanoma skin cancers, and in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma or breast) unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required during the study period.
   4. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the Investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patient to receive protocol therapy.
3. Treatment with anticancer medications, investigational drugs, surgery and/or radiation within the following interval before the first administration of study drug:

   1. < 14 days for chemotherapy, targeted small-molecule therapy, surgical resection of lesions or radiation therapy (prior palliative radiotherapy must have been completed at least 14 days prior to study drug administration). A 1-week washout is permitted for palliative radiation to non-CNS disease with Sponsor approval.

      Note: The use of denosumab against osteoporosis is permitted.
   2. < 28 days for prior monoclonal antibody used for anticancer therapy with the exception of PD-1 pathway-targeted agents.
   3. < 28 days or 5 half-lives (whichever is longer) before the first dose for all other investigational study drugs or devices. For investigational agents with long half-lives (e.g., > 5 days), enrolment before the fifth half-life requires Medical Monitor approval.
4. Receiving an immune-suppressive based treatment for any reason (including chronic use of systemic corticosteroid at doses > 10 mg/day prednisone equivalent) within 14 days prior to the first dose of study treatment (see the exception for CNS lesions described in 2a). Use of inhaled or topical steroids or brief corticosteroid use for radiographic procedures or systemic corticosteroids ≤ 10 mg is permitted.
5. Have received a live vaccine within 30 days of planned start of study therapy.
6. Have not recovered from toxic effect(s) of prior therapy to ≤ Grade 1, other than alopecia or fatigue.
7. Known allergy or reaction to any component of either study drug or formulation components.
8. Currently breastfeeding.
9. Known alcohol or other substance abuse.
10. Laboratory and medical history parameters not within Protocol-defined range. Absolute neutrophil count < 1.5 × 109/L.

    1. Platelet count < 100 × 109/L.
    2. Haemoglobin < 8 g/dL (transfusion is acceptable to meet this criterion).
    3. Serum creatinine ≥ 1.5 × institutional ULN or measured or calculated creatinine clearance (glomerular filtration rate can also be used in place of creatinine or CrCl) < 50 mL/min for patients with creatinine levels > 1.5 × institutional ULN.
    4. Aspartate aminotransferase, ALT, and alkaline phosphatase (ALP) ≥ 2.5 × ULN. Note: Patients with 1) bone metastases and 2) no hepatic parenchymal metastases on screening radiographic examinations may enrol if the ALP is < 5 × ULN. Patients with 1) bone metastases and 2) hepatic parenchymal metastases on screening radiographic examinations may enrol if the ALP is < 5 × ULN only with Medical Monitor approval.
    5. Total bilirubin ≥ 1.5 × ULN are excluded unless direct bilirubin is ≤ ULN. If there is no institutional ULN, then direct bilirubin must be < 40% of total bilirubin to be eligible (except patients with Gilbert syndrome - see Note below)
    6. International normalized ratio or prothrombin time (PT) > 1.5 × ULN.
    7. Activated partial thromboplastin time (aPTT) > 1.5 × ULN.
    8. Evidence of acute infection of hepatitis B virus (HBV), hepatitis C virus (HCV) and HIV. Patients who are on stable antiviral therapy and/or asymptomatic are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events [Safety and Tolerability] | Adverse event assessment will be assessed by CTCAE v5.0, through study completion, an average of 1 year.
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Cmax | at Cycle 0 Day 1 (pre-dose and 1/2/3-4/6-8hrs post-dose), and predose for Cycle 0 Day 7, Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15 and from Cycle 2 onwards Day 1 and End of Treatment. Cycle 0 is 7 days and Cycle 1 and onwards is 28 days.
  Peak plasma concentration
Cmin | at Cycle 0 Day 1 (pre-dose and 1/2/3-4/6-8hrs post-dose), and predose for Cycle 0 Day 7, Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15 and from Cycle 2 onwards Day 1 and End of Treatment. Cycle 0 is 7 days and Cycle 1 and onwards is 28 days.
  Minimum observed plasma concentration
t½ | at Cycle 0 Day 1 (pre-dose and 1/2/3-4/6-8hrs post-dose), and predose for Cycle 0 Day 7, Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15 and from Cycle 2 onwards Day 1 and End of Treatment. Cycle 0 is 7 days and Cycle 1 and onwards is 28 days.
  Terminal elimination half-life
tmax | at Cycle 0 Day 1 (pre-dose and 1/2/3-4/6-8hrs post-dose), and predose for Cycle 0 Day 7, Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15 and from Cycle 2 onwards Day 1 and End of Treatment. Cycle 0 is 7 days and Cycle 1 and onwards is 28 days.
  Time of the maximum observed plasma concentration
AUC0-t | at Cycle 0 Day 1 (pre-dose and 1/2/3-4/6-8hrs post-dose), and predose for Cycle 0 Day 7, Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15 and from Cycle 2 onwards Day 1 and End of Treatment. Cycle 0 is 7 days and Cycle 1 and onwards is 28 days.
  Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
AUC0-∞ | at Cycle 0 Day 1 (pre-dose and 1/2/3-4/6-8hrs post-dose), and predose for Cycle 0 Day 7, Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15 and from Cycle 2 onwards Day 1 and End of Treatment. Cycle 0 is 7 days and Cycle 1 and onwards is 28 days.
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
BED | for an average of 6 months
  Define the biologically effective dose (BED) of IOA-289 based on available parameters
CA19-9 | for an average of 6 months
  Assess changes of CA19-9 levels compared to baseline
LPA | for an average of 6 months
  Determine the PD activity of IOA-289, incl levels of LPA
Preliminary efficacy | Imaging for RECIST assessment will start at C2D1 ±3 Days and repeated every 8 Weeks (56 ± 5Days) until disease progression.
  Document preliminary signs of clinical efficacy of IOA-289 when given in combination with gemcitabine/nab-paclitaxel (e.g. overall response rate [ORR], duration of response [DOR], disease control rate (DCR), progression-free survival [PFS], and overall survival [OS] using RECIST v1.1)
Overall response rate [ORR] | for an average of 6 months
  ORR defined as percentage of patients with a CR or PR based on appropriate radiographic imaging and consistent with RECIST 1.1
Disease control rate [DCR] | for an average of 6 months
  DCR is defined as the combined percentage of patients with radiographic CR, PR and SD at different time points
Duration of response [DOR] | for an average of 6 months
  DOR defined as time from first documented evidence of CR or PR until disease progression or death from any cause among patients who achieve objective response
Progression free survival [PFS] | for an average of 6 months
  PFS defined as the time from the date of the first dose of study treatment until the earliest date of disease progression as determined by radiographic disease assessment
Overall survival [OS] | for an average of 6 months
  OS defined as the time from the date of the first dose of study treatment until death from any cause.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (2):
  - UO Oncologia of Azienda Ospedaliera Universitaria Integrata di Verona, Verona, Verona
  - Medical Oncology and Immunotherapy Unit, University Hospital of Siena, Siena
- Beatson West of Scotland Cancer Center, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khasabova IA, Khasabov SG, Johns M, Juliette J, Zheng A, Morgan H, Flippen A, Allen K, Golovko MY, Golovko SA, Zhang W, Marti J, Cain D, Seybold VS, Simone DA. Exosome-associated lysophosphatidic acid signaling contributes to cancer pain. Pain. 2023 Dec 1;164(12):2684-2695. doi: 10.1097/j.pain.0000000000002967. Epub 2023 Jun 6. PMID 37278638